CLINICAL TRIAL: NCT03950336
Title: Influence of Prebiotics on Intestinal Permeability in First Degree Relatives of Crohn's Patients
Brief Title: Prebiotics and Diet to Reduce "Leaky" Gut in First Degree Relatives of Crohn's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00090125
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Healthy First Degree Relatives of Crohn's Disease Patients
Keywords: intestinal permeability; Crohn's Disease (CD); oligofructose-enriched inulin; prebiotics; n-3 polyunsaturated fatty acids (n-3 PUFA); intestinal microbiota
MeSH Terms: conditions — Crohn Disease | interventions — Prebiotics; maltodextrin

STUDY DESIGN:
Intervention Model Description: placebo-controlled parallel study with two simultaneous interventions
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blind placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotics + "Low n-6 PUFA Diet" (Other): A combination of beta-fructans (12g/day) and a diet with reduced intake of n-6 PUFAs and higher intake of n-3 PUFAs.
  Interventions: Dietary Supplement: Prebiotics; Other: Low n-6 PUFA Diet
- Placebo + "Control Diet". (Other): A combination of maltodextrin (5g/day) and a control diet following the guidelines of Canada's Food Guide.
  Interventions: Dietary Supplement: Maltodextrin; Other: Control Diet

INTERVENTIONS:
Dietary Supplement: Prebiotics — Oligofructose-enriched inulin [a combination of shorter chain oligofructose, Degree of Polymerisation (DP) 3 - 9 and longer chain inulin (DP ≥ 10), in a 50:50 ratio ± 10 %] 12 g/day for 6 weeks
  Other Names: Prebiotin
  Arms: Prebiotics + "Low n-6 PUFA Diet"
Other: Low n-6 PUFA Diet — The Mediterranean diet pattern (MDP) with increased n-3 PUFA, saturated fatty acids (SFA) and monounsaturated fatty acids (MUFA) and reduced n-6 PUFAs food intake will be adopted as suitable Low n-6 PUFA diet.
  Other Names: Mediterranean - based Diet
  Arms: Prebiotics + "Low n-6 PUFA Diet"
Dietary Supplement: Maltodextrin — Maltodextrin consists of D-glucose units connected in chains of variable length (DP 3-17). The glucose units are primarily linked with α(1→4) glycosidic bonds. Maltodextrin is easily hydrolyzed by the intestinal enzymes and thus does not have an effect on colonic microbiota. Maltodextrin (5 g/days for 6 weeks) will be used as a placebo for the prebiotic treatment
  Arms: Placebo + "Control Diet".
Other: Control Diet — Participants who will not be assigned to "Low n-6 PUFA diet" will be advised to follow the Canada's Food Guide recommendations ("Control diet"). As Canada's Food Guide Diet is also designed with the aim to support healthy eating and prevention of metabolic and chronic disorders, this diet may not be considered as a true comparator for the Low n-6 PUFA diet intervention.
  Other Names: Canada's Food Guide-based Diet
  Arms: Placebo + "Control Diet".

SUMMARY:
Crohn's disease (CD) is a recurring inflammation of the intestines. The etiology is unknown; however evidence suggests that it could be a combination of gut microbes, environmental factors and genetics. CD has a strong genetic component, with up to 12% of patients having familial history. The Western diet is also thought to increase the risk of developing CD. In addition up to 20% of healthy first-degree relatives (FRD) of CD patients have increased small intestinal permeability ("leaky gut"). Previous studies have also shown that the Western diet can affect the intestinal immune response and normal intestinal barrier function, as well as alter the gut microbiota. We are interested in looking into whether beneficial dietary fibers (prebiotics) in combination with a diet low in n-6 polyunsaturated fatty acids (PUFAs) and high in n-3 PUFAs can protect against the development of CD.

Prebiotics are carbohydrates that cannot be digested by human enzymes and instead feed the bacteria in the colon that can digest them. Prebiotics occur in different fruits and vegetables. They have been shown to improve health by positively changing the gut microbes and their metabolism.

The prebiotic we will be using are β-fructans. β-fructans have been shown to reduce "leaky gut" and positively impact the intestinal immune system in experimental models and healthy humans. Diet has been shown to affect the gut microbes, intestinal inflammation development and the activity of prebiotics. We hypothesize that β-fructans in combination with a diet low in n-6 PUFAs / high in n-3 PUFAs (similar to a Mediterranean diet) can reduce intestinal permeability ("leaky gut") in FDR of CD patients, associated with beneficial changes in the gut microbes.

Participants (FDR of CD patients; 40 total) will be randomized and receive either a 12 g/day dose of the prebiotic oligofructose-enriched inulin (Prebiotin), or placebo (maltodextrin), as well as a dietary intervention. In order to control the n-3 and n-6 PUFA intake, participants will receive nutritional counselling by a registered dietitian. The Mediterranean diet will have the low n-6 and high n-3 intake ("Low n-6 PUFA"). Participants in the control diet group will be advised to follow the Canada's Food Guide (CFG) recommendations. Thus, this placebo-controlled study will involve 2 intervention groups with 20 participants in each group: 1) Prebiotic + Low n-6 PUFA; 2) Placebo + CFG.

DETAILED DESCRIPTION:
1. Background:

   Crohn's disease (CD) is a chronic intestinal inflammation, affecting approximately 130,000 Canadians. Its incidence and prevalence is rising worldwide. The disease etiology is unknown; however its pathogenesis is thought to be mediated by commensal gut bacteria, affected by environmental factors in a genetically susceptible host. It is well established that susceptibility to CD has a strong genetic component with up to 12% of the patients having family history of inflammatory bowel disease (IBD). Genome-wide association studies (GWAS) have identified more than 230 single nucleotide polymorphisms (SNPs) associated with IBD. However the risk-associated SNPs seems to account for only a portion of the observed IBD heritability, as many healthy individuals and relatives of Crohn's patients who carry these risk alleles never develop disease.

   The gut microbiome, which is also implicated in the CD pathogenesis, also has a certain degree of inheritance. Up to a third of the intestinal bacteria are heritable, raising the possibility of specific host genetic variants shaping the individual variability in microbial profiles. A study with 582 healthy individuals found that a high genetic risk for IBD was associated with a decrease in the relative abundance of the butyrate-producing Roseburia. Diet independently can affect the gut microbiome in short- and long term. Population-based studies in IBD indicate strong association of high dietary intakes of total fats, n-6 polyunsaturated fatty acids (PUFAs) and meats with increased risk of IBD, while high intake of fruits and vegetables decrease that risk. Animal studies have described the mechanisms underlying the pathogenesis of high-fat diets in colitis, including decreased Paneth cell area and less production of antimicrobial peptides by Paneth cells in the small intestines; reduced goblet cell number and less secreted mucin by goblet cells in the small intestines; reduced levels of tight junction proteins as occludin in the ileum, further illustrated by increased small intestinal permeability; increased IL-6 secretion in colon; and finally expanded abundance of pathobionts, such as Atopobium and Proteobacteria in stool. This data suggests that a high-fat diet (as an example of Western diet) has significant effect on the intestinal immunity and barrier function together with induction of dysbiosis and pathobiont expansion that can finally predispose to the development of inflammatory bowel disease.

   N-6 PUFAs have been identified as a risk factor for IBD. Canadians currently consume 5-10% dietary energy from n-6 PUFA, due to increased consumption of vegetable oils recommended by Canada's Food Guide. Meanwhile consumption of n-3 PUFAs (docosahexaenoic acid and eicosapentaenoic acid) with anti-inflammatory actions, represent only 0.15% dietary energy. Both n-6 and n-3 PUFAs are precursors of eicosanoids that regulate inflammation but in polarizing means. N-6 PUFAs, promote the production of pro-inflammatory series 2 prostaglandins (like prostaglandin E2, PGE2), thromboxanes and series 4 leukotrienes and also exacerbated murine colitis in several models. In contrast, n-3 PUFAs have anti-inflammatory properties that lead to the series 3 PGE, series 5 leukotrienes, and resolvins, which reduce translocation of inflammatory mediators to the site of injury. However clinical studies have shown conflicting results on the use of fish oil as source of n-3 PUFAs in IBD. Previously it was shown that fish oil can cause enrichment with gut pathobionts, and worsened mortality during infectious colitis in mice when added to n-6 PUFA rich diet, but not if combined with other fatty acids, revealing the importance of the background diet. Therefore a diet with reduced n-6 PUFA but higher fibre intake is proposed to be protective in IBD.

   Increased small intestinal permeability or so called "leaky gut" has been associated with many chronic conditions as obesity, type 2 diabetes and IBD. Increased intestinal permeability is also one of the potential pathogenetic risk factors for CD identified in up to 20% of our 10 years' longitudinal study population of healthy first-degree relatives (FDR) of Crohn disease patients. Furthermore, certain diets such as high-fat, high-glucose or high-fructose diets can also cause barrier dysfunction and increase the gut permeability, thus increasing the risk of developing metabolic endotoxemia and chronic intestinal inflammation. In contrast, reducing small intestinal permeability attenuates experimental colitis. These findings suggest that reduction of the gut permeability may reduce the risk factors leading to development of CD in FDR of CD patients.

   Studies conducted with animal models and healthy volunteers described reduction of gut permeability following consumption of β-fructans. However, the prebiotics efficacy in experimental IBD is also dependent on the background diet composition. We recently found that β-fructans protective effect in HLA-B27 rat colitis is modulated by n-6 and n-3 PUFAs intake. These data highlight that β-fructan type prebiotics are beneficial, but also suggest that background dietary lipid composition can modulate clinical outcomes. Since most Canadians consume a high n-6 / low n-3 PUFAs diet we propose that a combination of fatty acids including n-3 PUFAs will overpower n-6 PUFAs effect on β-fructans and (further) improve clinical response.
2. Study Hypothesis and Aims:

Based on the β-fructans efficacy in reducing intestinal permeability and regulating gut immunity shown in experimental models and clinical studies with healthy participants as well as the effect of diet on gut microbiome, colitis development and prebiotics activity, we hypothesize that β-fructans in combination with high n-3 PUFAs/low n-6 PUFAs diet (similar to a Mediterranean diet) can reduce small intestinal permeability and prevent chronic intestinal inflammation in FDR of CD patients, associated with improved intestinal microbiota metabolism.

In order to fulfill this hypothesis the following aims are proposed:

1. To assess if oral administration of β-fructans and dietary changes can improve small intestinal permeability (measured by urinary excreted lactulose and mannitol) in those FDRs with abnormal permeability.
2. To assess which protective mechanisms are associated with the permeability changes such as alterations in circulating zonulin, glucagone-like peptide 2 (GLP-2) and plasma endotoxin, as well as changes in gut microbiota composition and short chain fatty acid production.
3. Study Design:

Participants (first degree relatives of CD patients; 40 total) will be randomized to receive either β-fructans (12 grams daily dose of Prebiotin®, oligofructose-enriched inulin in ratio 1:1, equivalent to Orafti®Synergy1, supplied by Jackson GI Medical), or placebo (digestible maltodextrin, 5 grams daily dose, isocaloric to 12 g/d Prebiotin®) as well as dietary intervention. In order to control n-3 and n-6 PUFAs intake, participants will receive nutritional counselling by a registered dietitian. The Mediterranean diet pattern (MDP) (also called below "Low n-6 PUFA diet") with increased n-3 PUFA, saturated fatty acids (SFA) and monounsaturated fatty acids (MUFA) and reduced n-6 PUFAs food intake will be adopted as suitable low n-6 PUFA diet. Participants who will not be assigned to "Low n-6 PUFA diet" will be advised to follow Canada's Food Guide recommendations ("Control diet"). Thus this placebo-controlled study will involve 2 intervention groups with 20 participants in each arm: 1) Prebiotin + "Low n-6 PUFA Diet"; 2) Placebo + Control Diet

The intestinal permeability will be evaluated using lactulose/mannitol ratio (at weeks 0 and 6), as well as serum/plasma markers for intestinal permeability including zonulin, glucagone-like peptide 2 (GLP-2) and lipopolysaccharides (LPS) (weeks 0 and 6). We will also study the effect of prebiotic product and diet on fecal microbiota composition and activity (as fecal short-chain fatty acids and bile acids) (weeks 0 and 6). Attention will also be paid to the safety and tolerability of these prebiotics in FDR using questionnaires related to adverse events/dyspepsia and gastrointestinal habits (weeks 0, 3, and 6).

Since diet is also part of the intervention study and thought to play role in the intestinal permeability and prebiotic activity, all participants will receive dietary counselling and will be expected to adhere to recommended diet. Long-term dietary intake correlates with the bacteria taxa in the individual, so is important to quantify this prior to the dietary intervention. Participants will complete the on-line version of the Canadian Diet History Questionnaire II (C-DHQ II) which is a food frequency questionnaire to assess their pre-study diet (habitual diet) over the past year. In order to assess compliance to the diets the participants will complete the Canadian adaptation of the Automated Self-Administered 24-hour (ASA24-Canada-2016) which is a validated 24 hours dietary recall. The research dietitian will review recalls and provide feedback to participants based on results - in order to support changes to the diets. Additionally, participants will complete the Mediterranean Dietary Serving Score (MDSS). The MDSS is a validated instrument used to measure MDP adherence based on the consumption of food servings and food groups. The ASA-24 and MDSS will be completed at 0, 3 and 6 weeks of the study.

The study will be for 6 weeks from baseline where study participants will receive prebiotics treatment or placebo (maltodextrin) in addition to dietary counselling and intervention.

Oral intake of oligofructose-enriched inulin in a rat model of colitis as well in ulcerative colitis (UC) patients was able to increase fecal bifidobacteria and increase potentially protective butyrate-producing bacteria and their butyrate production in the colon and to alter cytokine production in the colon to favour a more anti-inflammatory profile. In the current proposed study we will assess if such microbiota changes driven by prebiotics and diet will also be associated with reduction of small intestinal permeability in the healthy population at risk for CD development. We will therefore measure small intestinal permeability at the start and at the end of the study, as well as collect stool, blood/serum and urine specimen throughout the trial.

Increased small intestinal permeability can also be caused by some broadly used medications such as nonsteroidal anti-inflammatory drugs (NSAIDs) including aspirin and ibuprofen. Virtually all studies agree that all conventional NSAIDs increase intestinal permeability in the human within 24 h of ingestion and that this is equally evident when they are taken long term. In order to control for this confounding factor, we will exclude individuals who take NSAIDs on daily basis. In addition, we will request participants to stop taking NSAIDs 1 week before the screening permeability test.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 15 - 50;
* First degree relative (parent, sibling, child) of patient diagnosed with Crohn's disease;
* Agree not to use any dietary supplements, herbal treatments, probiotics, prebiotics or dietary therapies within 1 week of starting the trial and during the study;
* Willingness to keep current physical activity during study period;
* Ability to give valid informed consent
* For females of childbearing potential and sexually active, a negative pregnancy test at screening, baseline and end-of-study, and accord to use appropriate birth control method (hormonal contraceptives, intrauterine devices, vasectomy/tubal ligation, barrier methods (condom or diaphragm), double-barrier methods or abstinence) during study period.

Exclusion Criteria:

* Use of probiotic and prebiotic supplements, fish oil or NSAIDS, prescribed or over the counter in the last 1 week;
* Use of antibiotics in the last 2 months;
* Celiac disease (allergic reaction to wheat products), gluten intolerance/sensitivity;
* Diabetes or uncontrolled / unstable blood glucose levels;
* Having history or evidence of significant gastrointestinal dysfunction and Irritable Bowel Syndrome (IBS);
* Having an active gastrointestinal infection (confirmed by stool pathogen culture test and Clostridioides difficile test)
* Having history or evidence of blood and bleeding disorder;
* Having uncontrolled or unstable blood pressure;
* Having a significant chronic disorder such as immune disorders, organ transplant, severe cardiac disease, renal failure, severe pulmonary disease, severe psychiatric disorder;
* Alcohol or drug abuse;
* Pregnant or lactating;
* Not able to consent to the study.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Change in small intestinal permeability over 6 weeks | week 0 and week 6
  Lactulose mannitol ratio test will be used for in vivo assessment of intestinal permeability. Increased intestinal permeability is defined as a ratio of lactulose/mannitol 0.025 or more. Lactulose/mannitol ratio < 0.025 is considered as normal.

SECONDARY OUTCOMES:
Changes in serum/plasma markers for intestinal permeability | weeks 0 and 6
  Zonulin, glucagon like protein 2 (GLP-2) and lipopolysaccharides (LPS) are chosen as markers for intestinal permeability
Changes in fecal microbiota and their metabolic activity | weeks 0 and 6
  Assessment by 16S ribosomal DNA (rDNA) microbial sequencing; short-chain fatty acids and bile acids measurement
Participant compliance and tolerability | weeks 0, 3 and 6
  Assessment by structured questionnaires, package counting and adverse events monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Levinus Dieleman, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared outside the study team.